CLINICAL TRIAL: NCT06182176
Title: Evaluating the Effectiveness and Cost-effectiveness of Integrating Mass Drug Administration for Helminth Control With Seasonal Malaria Chemoprevention in Ghanaian Children
Brief Title: Effectiveness and Cost-effectiveness of Integrated Model for Malaria and Helminth Control
Acronym: MALHELMIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Kintampo Health Research Centre, Ghana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29839
Record Dates: First submitted 2023-12-05; First posted 2023-12-26 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-12

CONDITIONS: Malaria; Soil Transmitted Helminths; Schistosomiasis; Seasonal Malaria Chemoprevention; Mass Drug Administration With Anthelminthic Drugs
MeSH Terms: conditions — Malaria; Schistosomiasis | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SMC plus anthelminthics group (Experimental): Anthelminthic drugs (albendazole and praziquantel) will be administered 24 hours (on Day 0) before administration of the following SMC drugs: Sulphadoxine-pyrimethamine (SP) on Day 1 and Amodiaquine (AQ) daily on Days 1, 2 and 3.
  Interventions: Drug: Sulphadoxine-pyrimethamine and Amodiaquine
- SMC group (Active Comparator): Participants randomized into the control communities will receive Vitamin A and Zinc supplements as control drugs on Day 0. On Day 1, these participants will receive the SMC drug (Sulphadoxine-pyrimethamine) (SP) and Amodiaquine (AQ) daily on Days 1,2 and 3.
  Interventions: Drug: Sulphadoxine-pyrimethamine and Amodiaquine

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine and Amodiaquine — The intervention drugs are standard drugs approved by the World Health Organisation for the preventive treatment of malaria (sulphadoxine-pyrimethamine and amodiaquine), schistosomiasis (praziquantel) and soil-transmitted helminths (albendazole).
  Other Names: SPAQ

SUMMARY:
Malaria remains a major health problem, especially among children living in sub-Saharan Africa where more than 90% of the disease and deaths occur. Adding to this high burden among the children is the co-existence of parasitic worms in their intestines and urinary tract. The combined infection of malaria and parasitic worms in these children has additive adverse effects of anaemia, poor physical and cognitive development, and death. Existing control programmes for the parasitic worms are operating sub-optimally despite the 2012 London Declaration on Neglected Tropical Diseases (NTDs) of achieving 75% treatment coverage by 2020. On the other hand, a malaria prevention programme, called Seasonal Malaria Chemoprevention (SMC), introduced in the same year as the London Declaration on NTDs has achieved more than 75% treatment coverage and prevented 75-85% of cases of uncomplicated and severe malaria in children. The remarkable success of SMC has led to the recent WHO recommendation for its extension to other at-risk age groups and in highly seasonal malaria transmission settings outside the Sahel region. This encouraging development supports the need to explore the possibility of integrating helminth control programmes with other successful delivery platforms such as SMC. However, limited empirical evidence exists on an integrated approach that integrated the control of malaria and parasitic worms in a safe, acceptable, easy-to-deliver and effective manner.

To address this knowledge gap, the investigators conducted a randomised controlled trial in the first stage of this project to establish the feasibility and safety of integrating helminth control with SMC among Senegalese children. This second stage will assess the effectiveness and cost-effectiveness of using SMC platform to deliver deworming drugs to preschool and school-aged children living in communities where the burden of malaria and parasitic worms is high in central Ghana. One thousand, two hundred children aged 1-14 years will be randomly assigned equally to two study communities where antimalarial (SMC) drugs and deworming drugs will be administered in combination to the children living in one study community, and antimalarial (SMC) drugs alone will be delivered to the children living in the second study community. The effectiveness of the combined delivery will be determined by checking whether the combined antimalarial and deworming drugs prevent anaemia in the children who receive the combined drugs compared to the children who receive antimalarial drugs only. We will also determine the cost and cost-effectiveness of this approach by estimating the incremental cost savings due to cases of moderate and severe anaemia averted by giving antimalarial and deworming drugs together to the children. The findings of this study would provide evidence to boost public health recommendations for an integrated control of malaria and parasitic worms among children living in the poorest countries of the world. The findings may also reinforce the empirical evidence that the future direction of healthcare systems in developing countries should be comprehensive health management rather than vertical management of a single disease.

DETAILED DESCRIPTION:
This study has two components: effectiveness and cost-effectiveness components. The effectiveness study will be conducted in three stages. The first stage will focus on pre-intervention surveys in Kintampo North Municipal and Pru East district. This will be followed by an intervention stage which will be conducted in either Kintampo North or Pru East district, depending on which of these districts has a higher prevalence of malaria, STH and schistosoma infections. The third stage will be a post-intervention cross-sectional survey in the communities where the intervention study is conducted.

First stage: During community sensitisation and engagement meetings with parents and caregivers of potentially eligible children living in Kintampo North Municipal and Pru East district, the Kintampo Health Research Centre (KHRC) study team will explain the need for this study, using a simple picture to illustrate the integration of SMC and anthelminthic drugs; the study rationale and informed consent procedure, and the risks and benefits of allowing their children to participate in the study. After these meetings, an investigator from KHRC will identify parents/caregivers of potential child participants to explain the study further to them on an individual basis. The parents/caregivers will be given a copy of the participant information sheet. Parents/caregivers who feel that the study is appropriate for their child will be visited at home at a mutually agreed time. For logistical purposes, written informed consent will be obtained from a parent/caregiver one day before the planned start date of the pre-intervention survey in both districts, along with positive assent from children aged ≥ 7 years, where required. Following this, an investigator will provide a pre-labelled stool collection container to the parent/caregiver at this visit and encourage them to collect stool from their child and keep this safely for the research team who will visit them the following day. Subsequently, the investigator will confirm the parent/caregiver's willingness to allow their child's continued participation in the study and administer a purpose-designed electronic questionnaire to the parents/caregivers. The questionnaire will cover information such as socio-demographic data, health and residence characteristics, history of de-worming and malaria treatment. Height/length (cm) and weight (kg) of each child will be measured and anthropometric indices height-for-age, weight-for-age, weight-for-height, and body mass index, will be calculated using the WHO AnthroPlus software (www.who.int/growthref/tools/en/). The study villages will be mapped by recording each study participant's household global-positioning system (GPS) coordinates with a hand-held GPS device.

Following administration of the questionnaire, finger-prick blood samples will be collected from each child participant for thick and thin smear examination for malaria microscopy, and blood spot filter papers will be collected for DNA isolation and PCR amplification for species determination. Haemoglobin concentrations will be measured using the Haemocue® method. Freshly voided urine samples will also be collected from all study children. Urine filtration test will be used to quantify S. haemotobium, according to standard laboratory guidelines. Parallel testing for circulating cathodic antigens (CCA) will be used to complement the filtration test.

Stool samples will be collected to detect intestinal helminths. Duplicate Kato-Katz thick smears will be prepared from the stool samples and examined by experienced technicians using light microscopy to determine the egg counts for S. mansoni and STH. The number of eggs per slide will be used to obtain a measure of the number of helminth eggs per gram of faeces (EPG). The intensity of the helminth infection will be categorised according to standard guidelines. A multiplex PCR assay will also be used for simultaneous detection of mixed infections of helminths. Quality control will be performed by re-examining at least 10% of randomly selected blood slides, urine filters and Kato-Katz smears by an experienced independent laboratory scientist. Laboratory staff performing the analyses will be masked to the origin of the samples.

Intervention stage: The intervention stage will be implemented during SMC campaign in Bono East Region. Results obtained from the laboratory analysis of the blood, stool and urine samples collected from the children enrolled in the pre-intervention surveys in Kintampo North and Pru East districts will be used to determine which of the districts will host the intervention stage of the study. Given that the focus of this project is to evaluate the effectiveness of the integrated SMC-NTD control programmes, the intervention stage of the study will be conducted in the district with a higher prevalence of malaria, STH and schistosomiasis. Also, the intervention stage will be implemented in conjunction with the SMC providers in the selected district. The first day of starting the intervention stage (Day 0) will correspond to the day prior to the commencement of the first cycle of SMC in the selected district. On that day, the communities in the selected district will be randomised at the community level and stratified on the basis of the malaria and helminth prevalence (obtained from the pre-intervention surveys) into two groups at a 1:1 ratio to receive either combined SMC and anthelminthic drugs (intervention arm) or SMC drugs only (control arm). Given that 4-aminoquinoline drugs are reported to have antagonistic pharmacological interactions with praziquantel, the SMC partner drugs, amodiaquine AQ (a 4-aminoquinoline derivative) and sulphadoxine-pyrimethamine (SP) will not be administered with anthelminthic drugs (albendazole and praziquantel) on the same day in this study. Therefore, eligible children randomised into the intervention communities will receive albendazole and praziquantel on Day 0 and those randomised into the control communities will receive Vitamin A and Zinc supplements as control drugs. On the following day which corresponds to the start (Day 1) of the first SMC cycle, the children in the control and intervention communities will receive AQ and SP according to the WHO and Ghana SMC implementation guidelines. This will be followed on the second and third day of the SMC cycle with all study children in the two groups receiving AQ, in line with the SMC guidelines. All children irrespective of the study arms will undergo safety assessment.

Post-intervention stage: All child participants enrolled in the intervention study will be evaluated one month after the last course of SMC cycles, which corresponds to the end of malaria transmission season, to measure their haemoglobin concentration and to obtain a further blood film, dried blood spot, stool and urine samples, to test for malaria-helminth co-infections using parasitological methods such as microscopy, Kato-Katz, urine filtration test and improved diagnostic tools including molecular methods (qPCR), as described above.

Data collection for the cost and cost-effectiveness analyses: The incremental financial and economic costs of delivering the integrated SMC-anthelminthic drugs programme in the intervention stage of this study will be estimated from a health service (Ministry of Health and donor) perspective, compared to the counterfactual of giving SMC drugs alone. Financial cost data (including all direct expenditures on the trial including salaries) and economic costs (donated goods or services, such as time of salaried health workers) will be collected through reviews of project records and semi-structured key informant interviews (KIIs) at district, health facility and community health workers (CHW) levels. Detailed costs will be captured for disaggregated cost categories, including SMC and MDA drugs; drug supply chain; CHW delivery of doses; supervision; training; planning meetings; sensitisation; and supplies. Incremental costs required for the integrated delivery of anti-helminth MDA with SMC above what would be required for SMC delivery alone will be identified. The cost of diagnosis and treatment of moderate and severe anaemia from the health service perspective will be estimated using a combination of primary and secondary data. Cost per outpatient visit and cost per inpatient day (excluding diagnosis and treatment) will be obtained from existing data sources. Costs of diagnostic tests, medicines and provider time for treating cases of moderate and severe anaemia will be captured through KIIs with health staff at facilities providing outpatient and inpatient services in the study area. These parameters will be used to estimate incremental cost savings due to cases of moderate and severe anaemia averted by SMC plus MDA compared to SMC alone.

For the cost-effectiveness analysis (CEA), the main measure of the effects will be disability-adjusted life-years (DALYs) averted. DALYs combine mortality (years of life lost, YLLs) and morbidity (years lived with disability, YLDs) into a single measure of effect, allowing the impact of SMC + MDA to be compared with the impact of different types of health interventions. The effect measure used to calculate DALYs will be moderate and severe anaemia cases averted (where anaemia is the primary outcome for the CEA which is where the main incremental health benefit from co-delivery is expected), derived from unadjusted results of the trial, calculated on the basis of intention-to-treat. DALYs will be modelled using a 3% discount rate in the base case, no age weighting, standard DALY weights and life tables, and other secondary data (e.g. duration of an episode of anaemia). The CEA results will be expressed as an incremental cost-effectiveness ratio (ICER). The ICER is calculated as the difference in costs between MDA + SMC versus SMC alone, divided by the difference in effects between those strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children aged 1-14 years;
* Provision of written informed consent by the parent/caregiver and a positive assent by children aged ≥ 7 years (in line with legal regulations in Ghana);
* Willingness to provide finger prick blood samples, urine, and stool samples;
* Residence in the study area for at least the past six months and willingness to be available in the study area for follow-up about 6 months after enrolment

Exclusion Criteria:

* Acutely ill child at the time of the drug administration;
* A child whose parents/caregivers decline to provide consent;
* A known HIV-positive child receiving co-trimoxazole prophylaxis;
* A child who has received a dose of either Sulphadoxine-pyrimethamine (SP), amodiaquine (AQ), albendazole (ALB) or praziquantel (PZQ) during the previous six months.
* A child with a known allergy to any of SP, AQ, ALB or PZQ.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
Change in Haemoglobin (Hb) concentration measured by HemoCue® | On the day of inclusion, and post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Comparison of the pre- and post-intervention values of Hb concentration of study children

SECONDARY OUTCOMES:
Incidence of clinical malaria, defined as fever of >37.5C | Detected by passive case detection during the surveillance period, an average of 5 months after co-administration of the study medications
  History of fever in the preceding 48 hours, and a positive malaria blood film with a parasite density of >0 per µl
Change in prevalence of anaemia on the day of inclusion, and post-intervention at the end of malaria transmission season; anaemia will be defined as Hb less than 11 g/dL | On the day of inclusion, and post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Comparison of the pre- and post-intervention values of Hb concentration of study children
Incidence of solicited adverse events and adverse drug reactions | During a period of six consecutive days after co-administration of study medications
  Safety assessment to be related to the study medications
Prevalence of P.falciparum and helminth co-infection | On the day of inclusion, and post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Prevalence of malaria-helminth co-infection
Density of P.falciparum and helminth co-infection | On the day of inclusion, and post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Density of malaria-helminth co-infection

OTHER OUTCOMES:
The cost per child treated per year and the cost per anaemia case averted | At post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Calculation by a cost analysis of the cost per child treated per year and the cost per anaemia case averted
Estimates of incremental cost-effectiveness | At post-intervention at the end of malaria transmission season i.e. one month after the last SMC cycle.
  Estimation of the incremental cost-effectiveness of integrated SMC plus anthelminthic treatment vs SMC alone, in terms of incremental economic costs per disability adjusted life year (DALY) averted.

CONTACTS AND LOCATIONS:
Overall Officials: Kwaku Poku Asante, MD, MPH, PhD, Study Chair — Kintampo Health Research Centre, Ghana; Muhammed O AFOLABI, MD, MPH, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Dennis Adu-Gyasi, PhD, Study Director — Kintampo Health Research Centre, Ghana; Brian O Greenwood, MD, Study Director — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: Yes
We will share the summary results of this trial or a link to the summary results within the trial registration record within 12 months of the study completion date
Supporting Information: Study Protocol, CSR
Time Frame: Within 12 months of the study completion date
Access Criteria: Open access requests will be entertained, the decision will be made by the Principal Investigator, quality of the request will be reviewed before granting it